CLINICAL TRIAL: NCT00306605
Title: Emotional Experiences in Fathers of NICU Babies: A Comparison of Fathers in Medical and Surgical NICUs.
Brief Title: Emotional Experiences in Fathers of NICU Infants
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Collaborators: Alfred I. duPont Hospital for Children (Other)
Responsible Party: Principal Investigator, Amy Mackley, Amy Mackley, Christiana Care Health Services
Other Study IDs: 26047
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Stress; Depressive Symptomatology
Keywords: Emotional experiences; fathers; stress; depressive symptomatology; NICU; preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Questionnaire — Participants will be asked to complete a questionnaire 3 times throughout the first 5 weeks after their infant's birth / hospitalization

SUMMARY:
This study is designed to evaluate the emotional experiences of fathers who have preterm infants who are hospitalized in a (neonatal intensive care unit)NICU setting. In addition, we will compare the emotional responses experienced by father of surgical NICU babies and fathers of medical NICU babies.

Our primary hypothesis is that paternal stress levels will be lower for those fathers of infants who are hospitalized in a medical NICU compared with fathers of infants who are hospitalized in a surgical NICU.

Secondary hypotheses include: 1) Stress levels for fathers of hospitalized infants will decrease over time; 2) Depressive symptomatology modulates perceived stress in fathers of NICU infants.

DETAILED DESCRIPTION:
It is well known that birth and hospitalization of a preterm infant is stressful for parents. Numerous studies have evaluated emotional factors such as maternal stress, parental role alteration, and maternal depression. Researchers have also investigated both maternal and paternal emotional responses in relation to their infant being hospitalized in the NICU. Studies examining paternal response alone have received less research attention. To date, no studies have compared the emotional response of fathers of medical NICU babies and fathers of surgical NICU babies.

The purpose of this study is to evaluate and compare perceived paternal stress and depressive symptomatology in fathers of preterm medical and surgical infants. Fathers who agree to participate will be given a questionnaire that is comprised of two self-report tools. Together these tools should take approximately 15-20 minutes to complete. Fathers who participate will be asked to complete these tools at three different times throughout their infants' stay in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* consenting fathers who are English speaking
* fathers with preterm infants < 30 weeks gestation and who are likely to survive
* Infants who lack congenital or genetic abnormalities likely to be associated with significant neurodevelopmental handicaps.

Exclusion Criteria:

* There are no specific exclusion criteria.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Fathers of preterm infants who are hospitalized in a newborn intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Perceived paternal stress levels will be lower for those fathers of infants who are hospitalized in a medical NICU compared with fathers of infants who are hospitalized in a surgical NICU. | First 5 weeks of infant's life and / or hospitalization

SECONDARY OUTCOMES:
Stress levels for fathers of hospitalized infants will decrease over time. | Within the first 5 weeks of their infant's birth / hospitalization
Depressive symptomatology modulates perceived stress in fathers of infants in NICUs. | First 5 weeks after their infant's birth / hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Amy B. Mackley, MSN, RNC, Principal Investigator — Christiana Care Health Systems; Michael L. Spear, MD, Principal Investigator — Christiana Care Health Systems; A.I. duPont Hospital for Children; Robert G. Locke, DO, Principal Investigator — Christiana Care Health Systems; A.I. duPont Hospital for Children; Rachel Joseph, MSN, CCRN, Principal Investigator — Alfred I. duPont Hospital for Children
Locations (2):
- United States (2):
  - Christiana Hospital (Christiana Care Health Systems), Newark, Delaware
  - A.I. duPont Hospital for Children, Wilmington, Delaware

REFERENCES:
- [Background] Miles MS, Brunssen SH. Psychometric properties of the parental stressor scale: infant hospitalization. Adv Neonatal Care. 2003 Aug;3(4):189-96. doi: 10.1016/s1536-0903(03)00138-3. PMID 14502526